CLINICAL TRIAL: NCT05928143
Title: Assessment of the Levels of Pain and Discomfort Associated With Corticotomy-assisted Retraction of the Anterior Maxillary Teeth Using Two Different Corticotomy Techniques. A Randomized Controlled Clinical Trial.
Brief Title: Patient Outcomes Associated With Two Accelerated Method of Retraction of Upper Front Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-12-2023
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Class II Division 1 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional corticotomy (Active Comparator): In this group, the acceleration procedure will be performed by elevating flaps and doing the surgical intervention directly using surgical burs.
  Interventions: Procedure: Traditional corticotomy
- Flapless corticotomy (Experimental): In this group, the acceleration procedure will be performed without elevating flaps, and the surgical intervention will be performed using a special device.
  Interventions: Procedure: Flapless corticotomy

INTERVENTIONS:
Procedure: Traditional corticotomy — A flap covering the alveolar process will be elevated. Perforations will be done using surgical burs, and then the flap will be returned, and sutures will be performed.
  Arms: Traditional corticotomy
Procedure: Flapless corticotomy — Some incisions will be made in the mucosa of the alveolar process. Then these incisions will allow the working head of the piezotome to cut the bone in grooves. The whole procedure will not require flap elevation and replacement.
  Arms: Flapless corticotomy

SUMMARY:
This study aimed to evaluate the levels of pain, discomfort, and functional impairment associated with traditional corticotomy and flapless corticotomy in the retraction of upper anterior teeth.

40 patients requiring extraction of maxillary first premolars and maximum anchorage to retract the upper anterior teeth will participate in the study. They will be divided randomly into two groups: flapless corticotomy (20 patients) and traditional corticotomy (20 patients).

DETAILED DESCRIPTION:
A corticotomy is the cutting of the bone that involves cortical bone only, leaving intact the medullary vessels and periosteum. It offers an advantage to adult patients in reducing orthodontic treatment time. The definition of traditional corticotomy is: elevating full-thickness periodontal flaps from a coronal approach, and vertical corticotomies are made between the teeth extending from 2-3 mm apical of the alveolar crest to 2 mm beyond the tooth apices and connected by a horizontal corticotomy; this process is done on both the labial and palatal aspects.

The definition of flapless corticotomy is a minimally invasive version of corticotomy, using a piezotome to inflict bone injury. This technique entails labial and palatal interproximal piezoelectric micro-incisions into the cortical bone without reflecting periodontal flaps.

Before enrolling each subject into the study, they will be examined completely to determine the orthodontic treatment plan. The operator will inform them about the aim of the study and ask them to provide written informed consent.

Self-drilling titanium mini-implants (1.6mm diameter and 8mm length) will be used. they will be inserted between the maxillary second premolar and first molar at approximately 8-10mm above the archwires at the mucogingival junction and will be checked for primary stability (mechanical retention). Then the maxillary first premolar will be extracted. The maxillary arch will be leveled and aligned. The rectangular stainless steel archwires (0.019" × 0.025") with anterior 8mm height soldered hooks distal to the lateral incisors will be inserted.

The surgery will be carried out under local anesthesia. The traditional corticotomy will be handled by the same maxillofacial surgeon, and the flapless corticotomy will be handled by the same orthodontist.

For traditional corticotomy, incisions in the mesial aspect of one-second premolar to the mesial surface of the contralateral second premolar will be placed, and a full-thickness flap will be elevated 3 mm above the apical region of the tooth. piezoelectric under copious irrigation will make vertical and horizontal cuts (only cortical surface). The vertical cuts will be between the dental roots in the interdental cortical surfaces, stopping 2 mm short of the alveolar crest occlusally. The horizontal cut will connect the vertical cuts 2 mm beyond the root apex. These cuts will be performed from the mesial aspect one-second premolar to the mesial surface of the contralateral second premolar involving the anterior. Similarly, a palatal flap incision will be raised immediately for doing the same vertical and horizontal cuts in the superficial surface of the palatal bone.

For the flapless corticotomy, the depth of gingival tissue will be determined through bone sounding using a periodontal probe. A scalpel will be used to make the incisions through the gingiva, 4mm below the interdental papilla, to preserve the coronal attached gingiva. These vertical incisions will be placed from the mesial aspect of the one-second premolar to the mesial surface of the contralateral second premolar on the labial and palatal aspects of the maxilla through the gingiva and the underlying bone. A piezo-surgery knife will be used to create the cortical alveolar incisions to a depth of 1 mm within the cortical bone.

The surgical procedure will be performed, and (250-300) g force will be applied on each side (3-4 days) after corticotomy using two Nickle-Titanium (NiTi) springs attached between the mini-implants and the soldered hooks in a direction approximately parallel to the occlusal plane for conducting an en-masse retraction. The force level will be measured every 2 weeks after the corticotomy. Retraction will be stopped when a class I canine relationship is achieved, and a good incisor relationship will be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy patients
2. Class II Division 1 malocclusion :

   * Mild/moderate skeletal Class II (sagittal discrepancy angle ≤7)
   * Overjet ≤10
   * Normal or excessive facial height (Clinically and then cephalometrically assessed using these three angles: mandibular/cranial base angle, maxillary/mandibular plane angle, and facial axis angle)
   * Mild to moderate crowding ≤ 4
3. Permanent occlusion.
4. Existence of all the upper teeth (except third molars).
5. Good oral and periodontal health:

   * Probing depth < 4 mm
   * No radiographic evidence of bone loss.
   * Gingival index ≤ 1
   * Plaque index ≤ 1

Exclusion Criteria:

1. Medical problems that affect tooth movement (corticosteroid, nonsteroidal anti-inflammatory drugs (NSAIDs))
2. Presence of primary teeth in the maxillary arch
3. Missing permanent maxillary teeth (except third molars).
4. Poor oral hygiene or Current periodontal disease:

   * Probing depth ≥ 4 mm
   * radiographic evidence of bone loss
   * Gingival index > 1
   * Plaque index > 1
5. Previous orthodontic treatment

Ages: 17 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Change in the levels of pain | After 24 hours of the surgical intervention; 4 days; 7 days; 14 days; 28 days
  Patients will be asked this question about their feeling of pain (Item no 01): 'What is the degree of pain you have experienced?' A standardized questionnaire will be used to assess pain, discomfort, and functional impairment levels during the active phase of treatment. The patient will be asked to specify a point on the visual analog scale (VAS), a 100-mm horizontal line with two focal points at its beginning and end (0: there is no pain - 100: the worst pain). The score will be determined by measuring the distance from the beginning until the point identified by the patient.
Change in the levels of discomfort | After 24 hours of the surgical intervention; 4 days; 7 days; 14 days; 28 days
  Patients will be asked this question about their feeling of discomfort: 'What is the degree of discomfort you have experienced?' A standardized questionnaire will be used to assess pain, discomfort, and functional impairment levels during the active phase of treatment. The patient will be asked to specify a point on the visual analog scale (VAS), a 100-mm horizontal line with two focal points at its beginning and end (0: there is no discomfort- 100: the worst discomfort). The score will be determined by measuring the distance from the beginning until the point identified by the patient.
Change in the perception of swelling | After 24 hours of the surgical intervention; 4 days; 7 days; 14 days; 28 days
  Patients will be asked this question about their feeling of swelling: 'What is the degree of swelling you have experienced?' A standardized questionnaire will be used to assess pain, discomfort, and functional impairment levels during the active phase of treatment. The patient will be asked to specify a point on the visual analog scale (VAS), a 100-mm horizontal line with two focal points at its beginning and end (0: there is no swelling- 100: the worst swelling). The score will be determined by measuring the distance from the beginning until the point identified by the patient.
Change in the levels of chewing difficulty | After 24 hours of the surgical intervention; 4 days; 7 days; 14 days; 28 days
  'What is the degree of mastication difficulties you have experienced?' A standardized questionnaire will be used to assess pain, discomfort, and functional impairment levels during the active phase of treatment. The patient will be asked to specify a point on the visual analog scale (VAS), a 100-mm horizontal line with two focal points at its beginning and end (0: there is no difficulty- 100: too much difficulty). The score will be determined by measuring the distance from the beginning until the point identified by the patient.
Change in the levels of swallowing difficulty | After 24 hours of the surgical intervention; 4 days; 7 days; 14 days; 28 days
  Patients will be asked this question about their feeling of swallowing: 'What is the degree of swallowing difficulties you have experienced?' A standardized questionnaire will be used to assess pain, discomfort, and functional impairment levels during the active phase of treatment. The patient will be asked to specify a point on the visual analog scale (VAS), a 100-mm horizontal line with two focal points at its beginning and end (0: there is no difficulty- 100: the worst difficulty). The score will be determined by measuring the distance from the beginning until the point identified by the patient.
Change in the levels of jaw movement restriction | After 24 hours of the surgical intervention; 4 days; 7 days; 14 days; 28 days
  Patients will be asked this question about their feeling about the jaw movement restriction: 'What is the degree of the jaw movement restriction you have experienced?' A standardized questionnaire will be used to assess pain, discomfort, and functional impairment levels during the active phase of treatment. The patient will be asked to specify a point on the visual analog scale (VAS), a 100-mm horizontal line with two focal points at its beginning and end (0: there is no restriction- 100: maximum restriction). The score will be determined by measuring the distance from the beginning until the point identified by the patient.
Level of satisfaction | This outcome will be assessed at 28 days following the surgical intervention
  Patients will be asked this question about their satisfaction level: 'What is your level of satisfaction on the orthodontic treatment provided?' A standardized questionnaire will be used to assess pain, discomfort, and functional impairment during the active phase of treatment. The patient will be asked to specify a point on the visual analog scale (VAS), a 100-mm horizontal line with two focal points at its beginning and end (0: there is no satisfaction- 100: the highest satisfaction). The score will be determined by measuring the distance from the beginning until the point identified by the patient.
The more discomfort procedure between two interventions | This outcome will be assessed at 28 days following the surgical intervention
  Patients will be asked this question: (Which surgical intervention was more discomfort ("extraction of premolars" or "the surgical procedure for acceleration"?) Assessment will be performed using a three-point scale: 1- premolar extraction, 2- surgical procedure, or 3-the same.
The willingness to undergo this procedure again | This outcome will be assessed at 28 days following the surgical intervention
  Patients would be asked this question about the possibility of repeating the surgical procedure if they had to make the decision again: 'Would you accept to undergo this treatment again?' Assessment will be performed using a two-point scale: Yes/No.

CONTACTS AND LOCATIONS:
Overall Officials: Hanin Khlef, DDS, MSc, Principal Investigator — Department of Orthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria
Locations (1):
- Orthodontics Department, Faculty of Dentistry, University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alfawal AMH, Hajeer MY, Ajaj MA, Hamadah O, Brad B, Latifeh Y. Evaluation of patient-centered outcomes associated with the acceleration of canine retraction by using minimally invasive surgical procedures: A randomized clinical controlled trial. Dent Med Probl. 2020 Jul-Sep;57(3):285-293. doi: 10.17219/dmp/120181. PMID 32909702
- [Background] Mousa MM, Hajeer MY, Burhan AS, Almahdi WH. Evaluation of patient-reported outcome measures (PROMs) during surgically-assisted acceleration of orthodontic treatment: a systematic review and meta-analysis. Eur J Orthod. 2022 Dec 1;44(6):622-635. doi: 10.1093/ejo/cjac038. PMID 35796046
- [Background] Charavet C, Lecloux G, Bruwier A, Rompen E, Maes N, Limme M, Lambert F. Localized Piezoelectric Alveolar Decortication for Orthodontic Treatment in Adults: A Randomized Controlled Trial. J Dent Res. 2016 Aug;95(9):1003-9. doi: 10.1177/0022034516645066. Epub 2016 Apr 29. PMID 27129491
- [Background] Lombardo L, Ortan YO, Gorgun O, Panza C, Scuzzo G, Siciliani G. Changes in the oral environment after placement of lingual and labial orthodontic appliances. Prog Orthod. 2013 Sep 11;14:28. doi: 10.1186/2196-1042-14-28. PMID 24326120
- [Background] Gibreal O, Hajeer MY, Brad B. Evaluation of the levels of pain and discomfort of piezocision-assisted flapless corticotomy when treating severely crowded lower anterior teeth: a single-center, randomized controlled clinical trial. BMC Oral Health. 2019 Apr 16;19(1):57. doi: 10.1186/s12903-019-0758-9. PMID 30991984